CLINICAL TRIAL: NCT07288502
Title: Adherence to Secondary Prevention Medications and Factors Influencing Adherence, After Acute Coronary Syndrome in Patient Attending a Tertiary Care Centre Of Nepal: A Descriptive Cross-sectional Study
Brief Title: Adherence to Secondary Prevention Drugs and Influencing Factors After Acute Coronary Syndrome in Patients at a Tertiary Center in Nepal
Status: Completed | Type: Observational
Sponsor: Institute of medicine, Maharagjung medical campus (Other)
Responsible Party: Principal Investigator, Abhishek Kumar Shah, Principal Investigator, Institute of medicine, Maharagjung medical campus
Other Study IDs: 290 (6-11) E2 081/ 082
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndromes (ACS); Adherence
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: My Experience of Taking Medicines (MYMEDS) questionnaire — This study does not involve a clinical or therapeutic intervention. Instead, it employs an assessment-based approach to evaluate medication adherence among post-Acute Coronary Syndrome (ACS) patients. The core instrument is the My Experience of Taking Medicines (MYMEDS) questionnaire, a validated, self-reported tool specifically designed to identify modifiable barriers to adherence in individuals prescribed secondary prevention medications. The questionnaire is structured into six sections that systematically explore patients' current medication use, their understanding and satisfaction with their prescribed regimen, specific concerns about the medicines, practical challenges in medication administration, difficulties in integrating medications into daily routines, and a detailed assessment of adherence to each individual secondary prevention drug over the preceding month. Utilizing primarily Likert-scale responses, the tool provides a nuanced understanding of adherence behaviors and t

SUMMARY:
This study aimed to assess adherence to secondary prevention medications among patients in Nepal following an Acute Coronary Syndrome (ACS) event and to identify factors affecting adherence. ACS was a major cause of morbidity and mortality globally and in Nepal, requiring effective secondary prevention to minimize recurrent cardiovascular events. However, adherence to prescribed medications remained low, especially in low- and middle-income countries like Nepal. Poor adherence could lead to increased healthcare burden, worsened patient outcomes, and higher mortality rates. To address this, the study evaluated patients' medication adherence through the MYMEDS questionnaire, a self-reported tool that was positively received for its simplicity and clarity. Conducted at the Manmohan Cardiothoracic Vascular and Transplant Centre in Nepal, the study involved a sample of adult patients who were readmitted or attending follow-ups post-ACS. The research gathered data on patient demographics, socioeconomic factors, clinical characteristics, and self-reported adherence barriers, analyzing these with SPSS to assess correlations with clinical outcomes.

The 12-month project consisted of phases for ethical approvals, data collection, analysis, and report dissemination. By identifying key barriers to adherence, the study aimed to inform targeted interventions that could enhance medication adherence, improve long-term cardiovascular outcomes, and reduce healthcare burdens in Nepal and other similar settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ACS, including ST-Elevation Myocardial Infarction (STEMI), Non-ST-Elevation Myocardial Infarction (NSTEMI), or Unstable Angina within the last 12 months
* Patients aged 18 years and older.
* Patients willing to participate and provide informed consent for the study.

Exclusion Criteria:

* Individuals who have not been diagnosed with ACS or those with other acute or chronic conditions that might influence medication adherence unrelated to ACS.
* Patients with cognitive impairments or mental health issues that prevent them from understanding or responding accurately to the study questionnaires.
* Patients with severe chronic conditions (e.g., terminal illness, advanced dementia) that may affect their ability to adhere to medication regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of adult patients (age ≥18 years) who have either come to OPD for follow-up or have been readmitted for having cardiac complications months after surviving ACS (including STEMI, NSTEMI, and unstable angina) in Manmohan Cardiothoracic Vascular and Transplant Centre, Nepal was selected via convenience sampling.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence to secondary prevention medications measured using the My Experience of Taking Medicines (MYMEDS) questionnaire | 1 year
  The primary outcome of this study is the level of adherence to prescribed secondary prevention medications among patients with Acute Coronary Syndrome (ACS). Medication adherence will be assessed using the My Experience of Taking Medicines (MYMEDS) questionnaire, a validated self-reported adherence assessment tool developed for patients prescribed secondary prevention medicines after myocardial infarction.
  Adherence will be specifically evaluated using Section 6 of the MYMEDS questionnaire, which assesses how frequently patients have taken each prescribed secondary prevention medication over the preceding one month. The medications assessed include antiplatelet agents, statins, beta-blockers, and angiotensin-converting enzyme inhibitors or angiotensin receptor blockers (ACE inhibitors/ARBs).
  Responses are recorded on a 5-point Likert scale:
  All of the time, Nearly all of the time, Most of the time, About half of the time, Less than half of the time.
  For the purpose of analysis, pat

SECONDARY OUTCOMES:
Patient-reported barriers to medication adherence assessed using the My Experience of Taking Medicines (MYMEDS) questionnaire | 1 year
  Secondary outcomes include the identification of patient-reported factors influencing adherence to secondary prevention medications. These factors will be assessed using Sections 2 to 5 of the MYMEDS questionnaire, which evaluate modifiable barriers to medication adherence.
  These sections assess:
  Patients' understanding of and satisfaction with prescribed medications
  Concerns and beliefs regarding potential harms or necessity of medicines
  Practical difficulties related to medication use (e.g., swallowing pills, opening containers, obtaining refills)
  Challenges in integrating medications into daily routines, including forgetfulness and inconvenience
  Responses are measured using a 4-point Likert scale (Strongly agree, Agree, Disagree, Strongly disagree).
  Higher agreement with barrier-related statements indicates greater perceived barriers to adherence.
  Results will be summarized as frequencies and proportions for each barrier domain.
Association between medication adherence and demographic and clinical factors | 1 year
  This outcome will assess the association between medication adherence status (adherent vs non-adherent) and patient demographic characteristics (age, sex, education level, occupation, place of residence, income) as well as clinical factors (type of ACS, comorbidities, and treatment received). This analysis aims to identify population subgroups at higher risk of non-adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Manmohan Cardiothoracic Vascular and Transplant Centre, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive clinical and sociodemographic information from a relatively small, identifiable group of ACS patients at a single tertiary centre, making robust de-identification difficult in the Nepali context. However, the aggregated findings, such as overall adherence pattern and analysis of demographic factors influencing adherence, will be presented in the final study report.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT07288502/Prot_SAP_ICF_000.pdf